CLINICAL TRIAL: NCT05171894
Title: A Multi-Center, Randomized, Double-Blind, Vehicle-Controlled, Sequential Group Comparison Study to Evaluate the Safety and Efficacy of Light Dose in Subjects With Port-wine Birthmarks Treated With Hemoporfin Photodynamic Therapy
Brief Title: A Study to Evaluate Efficacy and Safety of Light Dose in Subjects With PWB Treated With Hemoporfin PDT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Fudan-Zhangjiang Bio-Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: F0026-US201
Record Dates: First submitted 2021-11-15; First posted 2021-12-29 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Port-wine Birthmarks; Port-Wine Stain; Nevus Flammeus
Keywords: Hemoporfin; Port-wine Birthmarks; Port-Wine Stain; Nevus Flammeus; Photodynamic therapy
MeSH Terms: conditions — Port-Wine Stain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (6):
- Hemoporfin+A J/cm2 Green Light (Experimental): Participants will receive Hemoporfin 5 mg/kg of body weight via intravenous (IV) infusion and fixed laser irradiation for certain time.
  Interventions: Drug: Hemopfin+Green Light
- Hemoporfin+B J/cm2 Green Light (Experimental): Participants will receive Hemoporfin 5 mg/kg of body weight via intravenous (IV) infusion and fixed laser irradiation for certain time.
  Interventions: Drug: Hemopfin+Green Light
- Hemoporfin+C J/cm2 Green Light (Experimental): Participants will receive Hemoporfin 5 mg/kg of body weight via intravenous (IV) infusion and fixed laser irradiation for certain time.
  Interventions: Drug: Hemopfin+Green Light
- Placebo+A J/cm2 Green Light (Placebo Comparator): Participants will receive Vehicle (Saline) via intravenous (IV) infusion and fixed laser irradiation for certain time.
  Interventions: Device: Vehicle+Green Light
- Placebo+B J/cm2 Green Light (Placebo Comparator): Participants will receive Vehicle (Saline) via intravenous (IV) infusion and fixed laser irradiation for certain time.
  Interventions: Device: Vehicle+Green Light
- Placebo+C J/cm2 Green Light (Placebo Comparator): Participants will receive Vehicle (Saline) via intravenous (IV) infusion and fixed laser irradiation for certain time.
  Interventions: Device: Vehicle+Green Light

INTERVENTIONS:
Drug: Hemopfin+Green Light — All qualified subjects randomized to Hemoporfin PDT treatment to receive up to 3 cycles of treatment.
  Other Names: Hemopfin photodynamic therapy
  Arms: Hemoporfin+A J/cm2 Green Light; Hemoporfin+B J/cm2 Green Light; Hemoporfin+C J/cm2 Green Light
Device: Vehicle+Green Light — All qualified subjects randomized to vehicle PDT treatment to receive up to 3 cycles of treatment.
  Other Names: saline photodynamic therapy
  Arms: Placebo+A J/cm2 Green Light; Placebo+B J/cm2 Green Light; Placebo+C J/cm2 Green Light

SUMMARY:
This is a multi-center, randomized, double-blind, vehicle-controlled, and sequential group Phase 2 study. Eligible subjects aged 18 to 75 years old with PWB will receive Hemoporfin PDT or vehicle PDT in 8-week cycles at fixed drug dose (5 mg/kg) and different light fluence.

DETAILED DESCRIPTION:
This is a multi-center, randomized, double-blind, vehicle-controlled, and sequential group Phase 2 study. Eligible subjects aged 18 to 75 years old with PWB will receive Hemoporfin PDT or vehicle PDT in cycles at fixed drug dose (5 mg/kg) and different light fluences. This study will be conducted in two sequential stages, each contains the same schedule, which includes Screening Period, Treatment Period apart; subsequent treatment is based on efficacy evaluation, and End of Study.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be 18 to 75 years of age inclusive, at the time of signing the informed consent.
2. Subject is Fitzpatrick skin type I-VI.
3. A male subject must agree to use contraception during the Treatment Period and for at least 6 months after the last dose of study treatment and refrain from donating sperm during this period.
4. A female subject is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

   Not a woman of childbearing potential (WOCBP) . OR A WOCBP who agrees to follow the contraceptive guidance during the Treatment Period and for at least 30 days after the last dose of study treatment.
5. The subject has a clinical diagnosis of PWB located i) on the extremities, trunk, caudal cervical and/or retroauricular area (Stage One); ii) on the face and/or neck (Stage Two).
6. The longest diameter of the treatment area is ≥3 cm, and the short diameter is ≥2 cm.
7. Subject is capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.
8. Subject, in the Investigator's opinion, is in good general health and free of any disease state or physical condition that may impair the evaluation of PWB or expose the subject to an unacceptable risk by study participation.
9. If the subject has a history of epilepsy or seizure, the disease must remain stable for at least 6 months prior to C1D1.

Exclusion Criteria:

1. Subject is pregnant, lactating, or is planning to become pregnant during the study.
2. Subject has plaque/nodular changes and severe hypertrophy within the target PWB area.
3. Subject has Sturge-Weber syndrome.
4. Subject has any skin pathology or condition that, in the Investigator's opinion, could interfere with the evaluation of the study drug or requires use of interfering topical, systemic, or surgical therapy.
5. The subject has evidence of scarring within the target PWB area and/or the subject has a history of hypertrophic scarring or keloidal scarring.
6. Subject is immunosuppressed related to medication use and/or disease.
7. The subject has clinical abnormalities, as determined by the Investigator, which makes them unsuitable for receiving study treatment in the Investigator's opinion at Screening.
8. Subject has received any therapy on the treatment region that, in the Investigator's opinion, may affect the target PWB area.
9. Subject is known or in the opinion of the Investigator likely to be noncompliant with the requirements of the study protocol (eg, due to alcoholism, drug dependency, mental incapacity).
10. Subject has a history of either significant neurological events (such as major stroke) or a mental condition rendering him/her unable to understand the nature, scope, and possible consequences of the study.
11. Subject has an unstable cardiac disease or has any medical condition that in the opinion of the Investigator may worsen from receipt of study treatment or subject participation.
12. The subject has a history of cutaneous photosensitization, porphyria, or photodermatosis.
13. The subject has the need or has plans to be exposed to artificial tanning devices or excessive sunlight during the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2024-09-21 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Stage One：Incidence of any local and systemic adverse events. | From baseline until end of study, up to approximately 44 weeks
  To compare the efficacy of multiple light doses (fluence) of Hemoporfin PDT To investigate the safety of multiple light doses (fluence) of Hemoporfin/vehicle PDT in subjects with Port-wine birthmark (PWB) in the extremities, trunk, caudal cervical, and/or retroauricular area
Stage Two: Port Wine Birthmark-Investigator Global Assessment (PWB-IGA) scale score reduction. | From baseline until end of study, up to approximately 44 weeks
  To compare the efficacy of multiple light doses (fluence) of Hemoporfin PDT with vehicle PDT in subjects with PWB of face and/or neck.

SECONDARY OUTCOMES:
Stage One：Change from Baseline in overall PWB-IGA severity score and other scales. | From baseline until end of study, up to approximately 44 weeks
  To further evaluate the efficacy of multiple light doses (fluence) of Hemoporfin/vehicle PDT in subjects with PWB.
Stage Two: Change from Baseline in overall PWB-IGA severity score and other scales. | From baseline until end of study, up to approximately 44 weeks
  To further evaluate the efficacy of multiple light doses (fluence) of Hemoporfin/vehicle PDT in subjects with PWB.
Stage Two: Incidence of any local and systemic adverse events. | From baseline until end of study, up to approximately 44 weeks
  To investigate the safety of multiple light doses (fluence) of Hemoporfin/vehicle PDT in subjects with Port-wine birthmark (PWB)

OTHER OUTCOMES:
Stage One：Maximum observed plasma concentration (Cmax) of Hemoporfin | On the first day of the Cycle 1 (each cycle is 56 days)
  To check what time will it take to reach the maximum contraction of Hemoporfin
Stage One：Area under the concentration-time curve (AUC 0-∞) from time 0 to infinity of Hemoporfin | On the first day of the Cycle 1 (each cycle is 56 days)
  To check the drug profile for absorption, distribution, metabolism and excretion for Hemoporfin
Stage One：Terminal elimination half-life (t1/2) of Hemoporfin | On the first day of the Cycle 1 (each cycle is 56 days)
  To check how much time Hemoporfin will take to eliminate half of it's concentration from participants.
Stage One：Time to Cmax (Tmax) of Hemoporfin | On the first day of the Cycle 1 (each cycle is 56 days)
  To check what will be the maximum concentration participants will obtained of Hemoporfin

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - UCI Health Beckman Laser Institute & Medical Clinic, Irvine, California
  - Dermatology Cosmetic Associates of La Jolla, Inc. d/b/a West Dermatology Research Center, San Diego, California
  - Miami Dermatology and Laser Institute, Miami, Florida
  - Maryland Dermatology, Laser, Skin & Vein Institute, Hunt Valley, Maryland
  - St. Luke's University Health Network, Bethlehem, Pennsylvania